CLINICAL TRIAL: NCT01464632
Title: Prospective, Open Label Study of the Short-and Midterm Safety and Efficacy of the EPIK Uni-Compartmental Knee System in Community Practice
Brief Title: Post-Market Study of the EPIK Knee System
Acronym: EPIK
Status: Withdrawn | Type: Observational
Why Stopped: Unable to enroll any study participants.
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Sponsor
Other Study IDs: PS-707
Record Dates: First submitted 2011-11-02; First posted 2011-11-03 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis; Post Traumatic Degenerative Disease
Keywords: medial knee replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary: Post Market Study
  Interventions: Device: EPIK™ uni-compartmental knee

INTERVENTIONS:
Device: EPIK™ uni-compartmental knee — This device is intended for partial replacement of the articulating surfaces of the knee when only one side of the joint is affected due to compartmental primary degenerative or post-traumatic degenerative disease, previous tibial condyle or plateau fractures, deformity, or revision of previous arthroplasty.
  Other Names: EPIK

SUMMARY:
The purpose of this study is to determine the short-term (2 yr) and midterm (5 yr) cumulative revision rates of the EPIK™ Uni-compartmental Knee System.

DETAILED DESCRIPTION:
Medial uni-compartmental knee replacement (UKA) has been used for over 40 years to treat osteoarthritis (OA) of the knee. It is becoming more widely accepted as a treatment for early stage OA of the knee in order to preserve bony and ligamentous structures. The majority of the subjects who have received this knee are older (over 65 yrs) however, it is being used increasingly more frequently in younger individuals who have uni-compartmental knee disease so that bone may be spared in case the need arises in the future for a total knee arthroplasty. The study will take place at two sites within the United States and be managed by the Clinical Affairs Department at DJO Surgical in Austin, TX. The study will include only subjects who meet the indications for use criteria for the EPIK™ Uni-compartmental Knee System and who are candidates for UKA. Investigators will enroll up to 60 subjects at each of 2 sites within the United States, for a total of 100 subjects maximum.

ELIGIBILITY:
Inclusion Criteria:

* Meet the indications for use of the EPIK Uni-compartmental knee system
* Must be a primary surgery
* Have a primary diagnosis of OA in the medial knee compartment
* Have active and passive flexion > 90º
* Have a fixed flexion contracture < 10º
* Have an intact ACL and PCL
* Be a primary, unilateral surgery
* Have BMI ≤ 35.00
* Must not have infection (or history of infection within last 3 months), chronic or acute, local or systemic
* Must not be pregnant
* Be willing and able to sign the informed consent
* Be willing to follow study procedures, including all follow up visits
* Be over 18 years of age (≥ 18) and 60 years or younger (≤ 60) at time of consent

Exclusion Criteria:

* Prior total or uni-knee arthroplasty (must be a primary surgery)
* Patello-femoral joint symptoms
* Bilateral surgical procedures
* BMI > 35.00
* Muscular, neurological or vascular deficiencies which compromise the affected extremity
* Insufficient bone quality which may affect the stability of the implant
* Infection (or history of infection within last 3 months), chronic or acute, local or systemic
* Is younger than 18 years of age (<18) or over 60 (>60) years of age
* Mental conditions that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements
* High levels of physical activity (ex. Competitive sports, heavy physical labor)
* Documented (active) alcohol or drug addictions
* Loss of ligamentous structures
* Prisoner
* Metals sensitivity
* Subject is pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who are between 18 years of age and 60 years of age at time of consent and have one side of the knee joint affected by compartmental primary degenerative or post-traumatic degenerative disease, previous tibial condyle or plateau fractures or deformity.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Revision Rate Post Surgery | 5 years
  To determine the number of revisions that occur to total knee replacements after receiving the uni-compartmental knee replaceement.

SECONDARY OUTCOMES:
Revision rate post surgery | 2 year
  To determine the number of revisions that occur to total knee replacements after receiving the uni-compartmental knee replaceement.

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Sheely, D.O., Principal Investigator — Hill Country Sports Medicine
Locations (1):
- Hill Country Sports Medicine, Kyle, Texas, United States